CLINICAL TRIAL: NCT06219642
Title: Mindfulness Intervention Using Virtual Reality in Older Adults With Symptoms of Anxiety and Depression in Ecuador
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad San Francisco de Quito (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Ana F Trueba, Researcher, Universidad San Francisco de Quito
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-034M
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Symptoms of Depression and Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR mindfulness intervention (Experimental): The intervention consists of a total of 10 sessions each lasting 30 minutes. In each session, we fit participants with the VR headset with a smartphone running the Sites for VR app. The phone, placed in the viewing compartment of the headset, shows a nature scene of the participant's choosing. Once participants have acclimated to the scene and understand how to look around the VR scene (by moving their heads in different directions), we will read a mindfulness script with a guided body scan and instructions to engage participants through experiencing the virtual reality nature scene with all senses.
  Interventions: Behavioral: Mindfulness using virtual reality
- Phone call check-in (No Intervention): Investigators will call patients every week and ask how they are doing.

INTERVENTIONS:
Behavioral: Mindfulness using virtual reality — In each session, participants will be led through the following mindfulness script while using the VR device here is an abbreviated version with excerpts:
  "Look around. Try to bring yourself to the moment you are in. Notice the presence of the scene around you. How does the air feel against your skin?" "How do your feet feel against the ground? Where are you? What do you see?" "Do you hear anything?" "What do you smell? What do you taste? While you stay seated, imagine you are walking." "What body sensations are you experiencing? What thoughts are you having? What emotions are you feeling?" At the end of the intervention, participants are asked questions like, "What did you notice about your thoughts and mood before, during, and after the VR session? Did you notice a change in how your body felt or your emotions? Was there anything difficult or uncomfortable about the experience that you feel comfortable sharing?"
  Arms: VR mindfulness intervention

SUMMARY:
The availability of affordable hardware and rapidly growing content that can be freely accessed in the public domain raises the possibility of VR being used across the world globally and, in a very broad range of settings, including low-income populations and middle-income countries. The goal of this study is implement a randomized control trial using a low-cost VR mindfulness intervention within older adults in Quito, Ecuador compared. The control group will only receive a check-in phone call.

DETAILED DESCRIPTION:
We created a guided mindfulness intervention using low-cost VR (smartphones and Destek V5 headsets) for older adults with anxiety in Quito, Ecuador. This project is a collaboration between the Technology and Aging Lab at McLean Hospital and the Universidad San Francisco de Quito in Ecuador. Our goal is to recruit 90 older adults with anxiety from various outpatient settings in Quito. They will be randomized to control or to the intervention group. The control group gets a phone call in which they are asked how they are doing during 10 weeks. Those in the intervention group will receive 10 sessions of mindfulness using VR. We will use the free "Sites in VR" app and select different nature scenes for each intervention. The intervention consists of a total of 10 sessions each lasting 30 minutes. In each session, we fit participants with the VR headset with a smartphone running the Sites for VR app. The phone, placed in the viewing compartment of the headset, shows a nature scene of the participant's choosing. Once participants have acclimated to the scene and understand how to look around the VR scene (by moving their heads in different directions), we will read a mindfulness script with a guided body scan and instructions to engage participants through experiencing the virtual reality nature scene with all senses. The Ecuador team was trained by the McLean Team on the specifications of the intervention, to review the protocol, and to resolve any problems encountered during the administration of the intervention. The mindfulness sessions will be recorded with video and audio for quality control and intervention supervision to ensure that there is consistency in how the intervention is implemented.

ELIGIBILITY:
Inclusion Criteria:

* Normal cognitive functioning or mild cognitive impairment determined using the Montreal Cognitive Assessment (MoCA), being able to give written consent, and being a Spanish speaker. Exclusion criteria were

Exclusion Criteria:

* moderate to severe cognitive impairment, blindness or severe vision problems, deafness or hearing problems, history of dizziness, and current psychosis or mania.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Behavioral Activation Scale for Depression (BADS) | pre and 10 week post intervention
  Overall behavior activation
Mindfulness Attention Awareness Scale (MAAS) | pre and 10 week post intervention
  Mindfulness skills and state
Geriatric Depression Scale (GDS-15) | pre and 10 week post intervention
  depression symptoms
Generalized Anxiety Disorder (GAD-7) | pre and 10 week post intervention
  Anxiety symptoms

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | pre and 10 week post intervention
  Stress measure

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad San Francisco de Quito, Quito, Pichincha, Ecuador

IPD SHARING:
Plan to Share IPD: Yes
We can share analytical plan and outcome, as well as study protocol and informed consent to any researcher that requests it.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available during the process of publication if peer-reviewers would like to review it and post publication upon request
Access Criteria: Data is available upon request